CLINICAL TRIAL: NCT01046552
Title: Preoperative Versus Intraoperative Endoscopic Sphincterotomy for Management of Choledocholithiasis and Cholecystolithiasis
Brief Title: Comparison Between Pre and Intraoperative ERCP in Treatment of Common Bile Duct Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: ahmed abdel-raouf el-geidie, gastroenterology surgical center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ERCP123
Record Dates: First submitted 2010-01-05; First posted 2010-01-12 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2009-09

CONDITIONS: Common Bile Duct Stones.
Keywords: Choledocholithias; Common bile duct stones; Endoscopic retrograde cholangiopancreatography; endoscopic sphincterotomy; Preoperative; intraoperative; Laparoscopic common bile duct exploration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PES/LC (Active Comparator): preoperative ES followed by LC within the same hospital admission
  Interventions: Procedure: preoperative ERCP and LC
- LC/IOES (Active Comparator): laparoscopic cholecystectomy with intraoperative ercp under the same anesthesia
  Interventions: Procedure: Intraoperative ERCP and LC

INTERVENTIONS:
Procedure: preoperative ERCP and LC — preoperative ERCP followed by LC
  Arms: PES/LC
Procedure: Intraoperative ERCP and LC — LC and intraoperative ERCP
  Arms: LC/IOES

SUMMARY:
ERCP plays an important role in management of common bile duct stones. Herein the investigators compare preoperative against intraoperative ERCP.

210 were included but only 198 patients were randomly divided into two groups; PES/LC (100 patients) and LC/IOES (98 patients).

The total hospital stay were significantly shorter in the group of LC/IOES

ELIGIBILITY:
Inclusion Criteria:

* patients with gallstones and common bile duct stones

Exclusion Criteria:

* contraindications to ercp

contraindication to laparoscopy

biliary pancreatitis

refusal to participate

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2006-06; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
clearance of stones from the common bile duct | 6 months

SECONDARY OUTCOMES:
bile duct injuries, retained stones, hospital stay, surgical time, conversion to open cholecystectomy | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abdel-Raouf El-Geidie, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- See also: mansoura university — http://www.mans.edu.eg